CLINICAL TRIAL: NCT06181318
Title: Predicting the Outcomes of LIVEr Resection Using Quantitative Magnetic Resonance Imaging: the POLIVER Study
Brief Title: Quantitative MRI and Outcomes of Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Arianeb Mehrabi, MD, Professor Dr. med., Fundacao Champalimaud
Other Study IDs: POLIVER20230628
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Liver Cancer; Liver Failure; Bile Leak; Liver Metastases
Keywords: Liver surgery; Major hepatectomy; Posthepatectomy liver failure; Future liver remnant; quantitative multiparametric MRI
MeSH Terms: conditions — Liver Neoplasms; Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Participants will be recruited after they have been diagnosed and their treatment has been planned by a multidisciplinary tumor board. Patients indicated to undergo major liver resection (> 3 segments based on Brisbane classification [23]) will be eligible for participation.
  Interventions: Diagnostic Test: Multiparametric MRI scan of the liver

INTERVENTIONS:
Diagnostic Test: Multiparametric MRI scan of the liver — MRI scans will be performed at the Champalimaud Foundation using a 1.5T scanner after patients have fasted for 4 hours. Transverse abdominal T1 maps will be acquired to estimate extracellular fluid (which increases in cases of fibrosis and inflammation) and T2* maps will be acquired to estimate liver iron levels. These quantitative MRI maps will be laid onto the volumetric images of Couinaud segments. Multi-slice quantitative maps will be generated using Liver MultiScan software (Perspectum, UK) with operators blinded to patient status. T1 measurements will be adjusted for the iron level to give iron-corrected T1 maps (cT1). Reference ranges for cT1 have been defined in the general population. PDFF maps of the liver will be calculated using MRI multi-echo and spoiled-gradient-echo acquisition. No intravenous contrast agents will be used in Liver MultiScan maps and the total scan duration will be approximately 30 minutes.

SUMMARY:
The present observational study aims to assess the benefit of this quantitative multiparametric magnetic resonance imaging (MRI) in clinical practice, to quantify future liver remnant performance, and to accurately predict the risk of liver failure after major hepatectomy, among patients undergoing major liver resection.

The main questions to be answered are:

* Can multiparametric MRI predict the postoperative liver function?
* Can multiparametric MRI predict the postoperative liver-specific complications as well as mortality? With ethical approval and fully informed consent, patients being considered for major liver resection will undergo clinical assessment, blood sampling, and multiparametric MRI before surgery. For the primary outcome, 33 participants will be needed to detect a minimum correlation coefficient of 0.2 with 5% significance and 80% power.

DETAILED DESCRIPTION:
In patients being considered for major liver resection, volumetric and functional evaluation of the future liver remnant should ideally be combined to reduce the risk of posthepatectomy liver failure (PHLF) and other adverse outcomes. Quantitative multiparametric magnetic resonance imaging (MRI) can measure liver health by assessing parenchyma fibrosis and inflammation. This has shown promising results in predicting postoperative liver performance. The current study aims to assess the benefit of this MRI-based technology in clinical practice, to quantify future liver remnant performance, and to accurately predict the risk of liver failure after major hepatectomy.

Prospective observational clinical study in a single hepatobiliary surgery center. With ethical approval and fully informed consent, patients being considered for major liver resection will undergo clinical assessment, blood sampling, and multiparametric MRI before surgery. Postoperative liver function and complications will be reported for 90 days after surgery. Preoperative MRI assessment scores and postoperative outcomes will be correlated to determine whether multiparametric MRI scans can accurately predict the risk of postoperative liver-specific complications (primary endpoint) as well as postoperative liver function, surgery-specific complications, the overall complication rate, quality of hospital care, and length of stay. For the primary outcome, 33 participants will be needed to detect a minimum correlation coefficient of 0.2 with 5% significance and 80% power. This study will include 33 patients and results are expected in 2024. If successful, this investigation will support the use of quantitative multiparametric MRI to guide surgical decision-making. This will represent a non-invasive, diagnostic, volumetric, and segmental functional test for the preoperative workup of patients being considered for major hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) patients with an indication for elective major liver resection.
* Any benign or malignant indication.
* Provision of informed consent.
* MRI scan performed ≤ 7 days before surgery

Exclusion Criteria:

* Previous liver resection.
* Previous volume-enhancing procedures, such as portal vein embolization.
* Previous microwave ablation of liver lesions.
* Contraindication and/or inability to undergo contrast-enhanced MRI scan (including implanted metallic devices or foreign bodies, claustrophobia and contraindication for Primovist® administration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited after they have been diagnosed and their treatment has been planned by a multidisciplinary tumor board. Patients indicated to undergo major liver resection (> 3 segments based on Brisbane classification) will be eligible for participation. No change in treatment or intervention is proposed in the present study. All evaluations and analyses will take place at Champalimaud Clinical Centre. Patients who are being considered for major liver resection and have given informed consent will undergo a preoperative assessment, during which baseline clinical data and blood samples will be collected and a multiparametric MRI scan of the liver will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Predicting the posthepatectomy liver failure after major liver resection | 90 days postoperative
  Correlation between future liver remnant performance (combined measure of liver volume, PDFF, and cT1) and posthepatectomy liver failure after major liver resection
Predicting the posthepatectomy biliary leakage after major liver resection | 90 days postoperative
  Correlation between future liver remnant performance (combined measure of liver volume, PDFF, and cT1) and posthepatectomy biliary leakage after major liver resection
Predicting the posthepatectomy hemorrhage after major liver resection | 90 days postoperative
  Correlation between future liver remnant performance (combined measure of liver volume, PDFF, and cT1) and posthepatectomy hemorrhage after major liver resection

SECONDARY OUTCOMES:
Correlation between remnant liver function after major liver resection and incidence of major complications | 90 days postoperative
  Correlation between future liver remnant performance (combined measure of liver volume, PDFF, and cT1) and major complications according to Clavien-Dindo classification (>IIIA) after major liver resection
Correlation between remnant liver function after major liver resection and postoperative mortality | 90 days postoperative
  Correlation between future liver remnant performance (combined measure of liver volume, PDFF, and cT1) and mortality according to Clavien-Dindo classification (>IIIA) after major liver resection

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, the data generated by the current research that supports our future article, would be made available as soon as possible, wherever legally and ethically possible.
Supporting Information: Study Protocol, SAP, ICF